CLINICAL TRIAL: NCT03921580
Title: Pilot Study to Evaluate the Satiating Effect of Enriched Canned Tuna With Fibre or Polyphenols in a Group of Healthy Overweight Subjects
Brief Title: Enriched Canned Tuna With Fibre or Polyphenols on Satiety
Acronym: SACIATUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Friobas Basilio S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 5048
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2018-06

CONDITIONS: Overweight
Keywords: Satiety; Polyphenols; Fibre; Visual Analogue Scale; Cross-over; Tuna
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Canned Tuna (Placebo Comparator): Control Canned Tuna
  Interventions: Other: Control Canned Tuna
- Enriched Canned Tuna Variety 1 (Experimental): Enriched Canned Tuna Variety 1: Wakame fiber
  Interventions: Other: Enriched Canned Tuna Variety 1
- Enriched Canned Tuna Variety 2 (Experimental): Enriched Canned Tuna Variety 2: Polyphenols
  Interventions: Other: Enriched Canned Tuna Variety 2

INTERVENTIONS:
Other: Control Canned Tuna — 210 g/day
  Arms: Control Canned Tuna
Other: Enriched Canned Tuna Variety 1 — 210 g/day
  Arms: Enriched Canned Tuna Variety 1
Other: Enriched Canned Tuna Variety 2 — 210 g/day
  Arms: Enriched Canned Tuna Variety 2

SUMMARY:
The purpose of this study is to evaluate the satiating effects of different canned tuna preserved in olive oil enriched with soluble fiber or polyphenols on overweight subjects (BMI ≥25 and <30 kg / m2).

Some studies have shown the contribution of high-fiber foods in the reduction of the cardiovascular risk.

DETAILED DESCRIPTION:
A randomized, cross-over and double-blind pilot study with 3 study arms is being performed to evaluate the satiating properties of different canned tuna preserved in olive oil enriched with soluble fiber or polyphenols on overweight subjects.

The investigators included 12 participants (6 men and 6 women) between 18 and 55 years (BMI ≥25 and <30 kg / m2). All volunteers will be randomized into 3 study groups, and participants will receive the 3 different study products in order during the 3 experimental phases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 65 years old.
* Body Mass Index (BMI) ≥25 and <30 kg/m2.
* Adequate cultural level and understanding for the clinical trial.
* Signed informed consent

Exclusion Criteria:

* Subjects with BMI ≥30 or <25 kg /m2
* Subjects diagnosed with Diabetes Mellitus.
* Subjects with dyslipidemia on pharmacological treatment
* Subjects with hypertension on pharmacological treatment
* Subjects with established diagnosis of eating disorder
* Smokers or those subjects with high alcohol consumption (> 2-3 servings/ day in men and> 1 serving/day in women (1 serving = 1 glass of wine or 1 bottle of beer)
* Subjects under pharmacological treatment (except oral contraceptives)
* Subjects with large weight fluctuations of more than 4 kg or who have undergone in six months a weight loss diet
* Subjects with sensory problems
* Subjects with gastrointestinal diseases that affect the digestion or absorption of nutrients
* Pregnant or breastfeeding women
* Women with menstrual irregularities (absence of menstrual cycle at least 2 months)
* Subjects with intense physical activity.
* Subjects with food allergies to meals included in breakfast, study product or lunch or that reject their consumption
* Subjects with a diagnosis of celiac disease or a gluten intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 6 men and 6 women
Enrollment: 12 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Satiety Hunger Assessment | Day 1, 8, 15
  Visual Analogue Scale (VAS). 100mm horizontal line anchored at each end with the extremes of the subjective feeling to be quantified. Subjects are instructed to rate the sensation being experienced according to how they define the line.
  e.g., "not at all hungry" (0mm) and "as hungry as I have ever felt" (100mm). Multiple measures are taken at repeated time intervals described below.

SECONDARY OUTCOMES:
Change from Baseline Blood Hormonal Satiety Markers | Day 1, 8, 15
  Concentration of Glucagon-like peptide-1 (GLP-1), Peptide tyrosine-tyrosine (YY), Ghrelin, Leptin, Ghrelin, Leptin, Gastric Inhibitory Peptide (GIP), Peptide C
Amount of food consumed in a "food ad libitum" | Day 1, 8, 15
  120 min After eating the study product
Total amount of food consumed in 24h | Day 1, 8, 15
  24h Food Record Method
Change from Baseline Glucose Metabolism Parameters | Day 1, 8, 15
  Concentration of Glucose
Change from Baseline Lipid Metabolism Parameters | Day 1, 8, 15
  Concentration of Cholesterol, LDL-C, HDL-C, TAG
Anthropometric Parameters | Day 1, 8, 15
  Weight and height will be combined to report BMI in kg/m2
Sensory Perception Test | Day 1, 8, 15
  Questionnaire of analysis of sensory perception of the food study product. Five questions that are valued on a scale of 0% to 100% asking about the taste and smell of the study product: desire with which the product is taken, taste, smell, consistency and what wait for effectiveness.
Adverse Effects | Day 1, 8, 15
  Number of participants gastrointestinal symptoms (Nausea, Diarrhea, Bloating and other disorders)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, MD, PhD, Principal Investigator — La Paz University Hospital
Locations (1):
- La Paz University Hospital, Madrid, Spain